CLINICAL TRIAL: NCT01503060
Title: Effectiveness of Parent-Led Interventions in Reducing Infant Hypersensitivity to Pain: A Longitudinal Randomized Controlled Trial
Brief Title: Effectiveness of Parent-Led Interventions in Reducing Infant Hypersensitivity to Pain
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Anna Taddio, Adjunct Scientist/Pharmacist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 1000025726
Record Dates: First submitted 2011-12-29; First posted 2012-01-02 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Pain
Keywords: pediatrics; Pain; Immunization
MeSH Terms: conditions — Pain | interventions — Water; Sucrose; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Placebo Comparator): * Visit 1-4 (2,4,6,12 month vaccinations): Patients will receive standard care
  * Visit 5 (15 month vaccination): At the last visit all 4 groups will receive all three active interventions.
  Interventions: Behavioral: Educational Video - Sham; Drug: Sucrose Placebo (water); Drug: Lidocaine Placebo
- Group 2 (Active Comparator): * Visit 1-4 (2,4,6,12 month vaccinations): Parents will be taught about managing pain
  * Visit 5 (15 month vaccination): At the last visit all 4 groups will receive all three active interventions.
  Interventions: Behavioral: Educational video - Active; Drug: Sucrose Placebo (water); Drug: Lidocaine Placebo
- Group 3 (Active Comparator): * Visit 1-4 (2,4,6,12 month vaccinations): Parents will be taught about managing pain and their infant will be given sugar
  * Visit 5 (15 month vaccination): At the last visit all 4 groups will receive all three active interventions.
  Interventions: Behavioral: Educational video - Active; Drug: Sucrose; Drug: Lidocaine Placebo
- Group 4 (Active Comparator): * Visit 1-4 (2,4,6,12 month vaccinations): Parents will be taught about managing pain and their infant will be given sugar water and a topical anesthetic
  * Visit 5 (15 month vaccination): At the last visit all 4 groups will receive all three active interventions.
  Interventions: Behavioral: Educational video - Active; Drug: Sucrose; Drug: Lidocaine

INTERVENTIONS:
Behavioral: Educational video - Active — The active video will instruct parents in techniques related to optimal infant soothing.
  Arms: Group 2; Group 3; Group 4
Behavioral: Educational Video - Sham — The sham video will provide general information about immunization immunization pain management.
  Arms: Group 1
Drug: Sucrose Placebo (water) — Infants will receive 2mL of liquid on the tongue 2 minutes prior to vaccination
  Arms: Group 1; Group 2
Drug: Sucrose — Infants will receive 2mL of liquid on the tongue 2 minutes prior to vaccination
  Arms: Group 3; Group 4
Drug: Lidocaine Placebo — Infants will receive 1 g of cream to one or both injection site(s), as required, for 20-30 minutes prior to vaccination
  Arms: Group 1; Group 2; Group 3
Drug: Lidocaine — Infants will receive 1 g of cream to one or both injection site(s), as required, for 20-30 minutes prior to vaccination
  Arms: Group 4

SUMMARY:
The aim of this study is to find out the effects of routinely using different types of pain-relieving strategies during routine immunization injections performed in infants.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants undergoing vaccination.

Exclusion Criteria:

1. preterm birth (<37 weeks gestation)
2. prior hospitalization/surgery (other than postnatal care),
3. documented/ suspected sensitivity/allergy to amide anaesthetics/vaccines,
4. mother plans to breastfeed or to use topical anesthetics or sugar water during injection.

Ages: 2 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 352 (Estimated)
Dates: Start 2011-12; Primary Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Hypersensitivity to pain | At 15 month vaccination (Visit 5)
  This will be assessed by comparing the pain scores between each active group and the placebo group at 15 months

SECONDARY OUTCOMES:
Effectiveness of interventions | At 2,4,6,12 month vaccinations (Visit 1-4)
  This will be assessed by comparing the pain scores between groups

CONTACTS AND LOCATIONS:
Overall Officials: Anna Taddio, PhD, Principal Investigator — The Hospital for Sick Children
Locations (2):
- Canada (2):
  - Outpatient Clinic, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

REFERENCES:
- [Derived] Taddio A, Riddell RP, Ipp M, Moss S, Baker S, Tolkin J, Dave M, Feerasta S, Govan P, Fletcher E, Wong H, McNair C, Mithal P, Stephens D. A Longitudinal Randomized Trial of the Effect of Consistent Pain Management for Infant Vaccinations on Future Vaccination Distress. J Pain. 2017 Sep;18(9):1060-1066. doi: 10.1016/j.jpain.2017.04.002. Epub 2017 Apr 26. PMID 28455250
- [Derived] Taddio A, Riddell RP, Ipp M, Moss S, Baker S, Tolkin J, Malini D, Feerasta S, Govan P, Fletcher E, Wong H, McNair C, Mithal P, Stephens D. Relative effectiveness of additive pain interventions during vaccination in infants. CMAJ. 2017 Feb 13;189(6):E227-E234. doi: 10.1503/cmaj.160542. Epub 2016 Dec 12. PMID 27956393